CLINICAL TRIAL: NCT05487209
Title: Clinical Value of the MRI Combined With SCC-Ag for the Diagnosis of High-grade Cervical Squamous Neoplasia (Cervical Intra-epithelial Neoplasia Grades 2 and 3 (CIN 2/3))
Brief Title: Clinical Value of the MRI Combined With SCC-Ag for the Diagnosis of HSIL (CIN 2/3)
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2022-07-204
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-08

CONDITIONS: Magnetic Resonance Imaging Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postmenopausal group
  Interventions: Diagnostic Test: MRI,SCC-Ag
- non-menopausal group
  Interventions: Diagnostic Test: MRI,SCC-Ag

INTERVENTIONS:
Diagnostic Test: MRI,SCC-Ag — Magnetic Resonance Imaging examination,serum squamous cells carcinoma antigen

SUMMARY:
The study aimed to identify the clinical value of Magnetic Resonance Imaging examination (MRI)combined with serum squamous cells carcinoma antigen (SCC-Ag) in women with high-grade squamous intraepithelial lesion (cervical intraepithelial neoplasia grades 2-3 (CIN 2-3)).

DETAILED DESCRIPTION:
186 female patients with the HSIL(CIN2-3) were included in this study and followed up from the time of admission. All patients underwent colposcopy examination, MRI, SCC-Ag, loop electrosurgical excision procedure (LEEP), extrafascial hysterectomy, or radical hysterectomy. Pathological findings of the patient's tissues were used as the final diagnostic criteria. On the one hand, we compared the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of MRI+SCC-Ag, LEEP of the menopausal group, and non-menopausal group. On the other hand, evaluating the accuracy of MRI combined with SCC-Ag examination in diagnosing HSIL(CIN2-3) by receiver-operating characteristic curve (ROC)．

ELIGIBILITY:
Inclusion Criteria:

* No previous history of cervical lesions
* TCT and HPV test results suspected cervical lesions
* Further colposcopy showed HSIL or CIN 2-3
* All selected patients underwent MRI, serological tests for SCC-Ag levels, LEEP, or radical hysterectomy

Exclusion Criteria:

* Patients with receiving cold knife conization
* Patients with skin squamous cell carcinoma or previous history of cancer
* Pregnant women
* Patients with serious heart, liver, kidney, blood system and autoimmune diseases

Ages: 26 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study conformed to the declaration of Helsinki and was approved by the Ethics Committee of Second Affiliated Hospital of Wenzhou Medical University. we prospectively collected the data of patients with HSIL(CIN2-3) from March 1 to September 31, 2021, all patients included in this study were followed up from admission to discharge. A total of 186 patients were eligible and signed written informed consent.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The number of cases whose combined diagnosis of MRI and SCC Ag In postmenopausal women | 20 days
  In postmenopausal women, the number of cases whose combined diagnosis of MRI and SCC Ag consistent with the final pathological results
the number of cases whose combined diagnosis of MRI and SCC Ag for the non-menopausal group. | 20 days
  In non-menopausal women, the number of cases whose combined diagnosis of MRI and SCC Ag consistent with the final pathological results

CONTACTS AND LOCATIONS:
Overall Officials: Zhao, Principal Investigator — The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU
Locations (1):
- The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Siegel RL, Ward EM, Jemal A. Global Cancer Incidence and Mortality Rates and Trends--An Update. Cancer Epidemiol Biomarkers Prev. 2016 Jan;25(1):16-27. doi: 10.1158/1055-9965.EPI-15-0578. Epub 2015 Dec 14. PMID 26667886
- [Background] Paavonen J, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Skinner SR, Hedrick J, Jaisamrarn U, Limson G, Garland S, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Jenkins D, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by oncogenic HPV types (PATRICIA): final analysis of a double-blind, randomised study in young women. Lancet. 2009 Jul 25;374(9686):301-14. doi: 10.1016/S0140-6736(09)61248-4. Epub 2009 Jul 6. PMID 19586656
- [Background] Fan A, Zhang L, Wang C, Wang Y, Han C, Xue F. Analysis of clinical factors correlated with the accuracy of colposcopically directed biopsy. Arch Gynecol Obstet. 2017 Nov;296(5):965-972. doi: 10.1007/s00404-017-4500-z. Epub 2017 Sep 9. PMID 28889237
- [Background] Sun X, Lei H, Xie X, Ruan G, An J, Sun P. Risk Factors for Residual Disease in Hysterectomy Specimens After Conization in Post-Menopausal Patients with Cervical Intraepithelial Neoplasia Grade 3. Int J Gen Med. 2020 Nov 10;13:1067-1074. doi: 10.2147/IJGM.S280576. eCollection 2020. PMID 33204141
- [Background] Chen P, Jiao L, Ren F, Wang DB. Clinical value of serum squamous cell carcinoma antigen levels in predicting chemosensitivity, lymph node metastasis, and prognosis in patients with cervical squamous cell carcinoma. BMC Cancer. 2020 May 14;20(1):423. doi: 10.1186/s12885-020-06934-x. PMID 32410650